CLINICAL TRIAL: NCT01567631
Title: Laparoscopic Anatomical Hepatectomy With Intrahepatic Glisson's Approach Versus Laparoscopic Anatomical Hepatectomy With Classical Procedure
Brief Title: Classical Procedure Versus Intrahepatic Glisson's Approach
Acronym: LAHIGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shuguo Zheng, MD (Other)
Responsible Party: Sponsor-Investigator, Shuguo Zheng, MD, Professor of Hepatobiliary Surgery Institute; Chief Physician; Administrator of laparoscopic department, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWHZSG002; Zhengshuguo (Registry Identifier: Zhengshuguo)
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Liver Diseases; Liver Neoplasms; Hepatic Haemangioma
Keywords: Classical Procedure; Intrahepatic Glisson's Approach; laparoscopic hepatectomy; Minimal invasive surgery; Endoscopic stapling devices
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intrahepatic Glisson's approach (Experimental)
  Interventions: Procedure: intrahepatic Glisson's approach
- classical hepatectomy (Active Comparator)
  Interventions: Procedure: classical hepatectomy

INTERVENTIONS:
Procedure: intrahepatic Glisson's approach — Forty patients with liver disease were selected and divided into intrahepatic Glission's group as described in the detailed description.Total laparoscopic hepatectomy with intrahepatic Glisson's approach were performed. Operation began with division of liver ligaments, liver mobilization, followed by intrahepatic access to the Glissonian pedicle (containing arterial, portal, and bile duct branches ). A endoscopic stapler devices was used for Glissonian pedicle cutting and suture. Liver parenchyma was divided by harmonic scalpel combined with vascular stapler. The specimen was extracted through suprapubic incision.
  Other Names: Laparoscopic with Intrahepatic Glssion's approach
  Arms: intrahepatic Glisson's approach
Procedure: classical hepatectomy — Forty patients with liver disease were selected and divided into classical laparoscopic hepatectomy group as described in the detailed description.Total laparoscopic anatomical hepatectomy with classical procedure were performed.The initial step is to dissect hepatic portal and expose the liver artery, portal Vein branch and the bile duct. Then endoscopic stapler devices were used to cut the canal mentioned above. Final step is to divide the liver parenchyma along the following ischemic delineation.
  Other Names: Laparoscopic anatomical hepatectomy with classical procedure
  Arms: classical hepatectomy

SUMMARY:
The purpose of this research is to compare the classical procedure with intrahepatic Glisson's approach for laparoscopic anatomical hepatectomy. The validity, feasibility and limitations were assessed objectively through our clinical prospective study. The investigators expect laparoscopic anatomical hepatectomy with intrahepatic Glisson's approach is safe, effective and feasible.

DETAILED DESCRIPTION:
Background: China is the high incidence area of liver disease, some of which need to be treated by surgical liver resection. The development of minimal invasive techniques opened up a new situation for hepatectomy. Intrahepatic Glisson's approach and the classical procedure are the two major operation procedures used in laparoscopic hepatectomy. The intrahepatic Glisson's approach has the advantages of less intraoperative bleeding and shorter operation time in our experience and as previous studies. The investigators expect further comparison of the safety and efficacy through this prospective controlled study by using two kinds of operation procedures.

Intervention: Classical procedure versus intrahepatic Glisson's approach: a prospective randomized study. Eighty patients with liver disease need undergo hepatectomy were selected and divided into intrahepatic Glisson's group and classical procedure group randomly, each group contains 40 cases. Total laparoscopic hepatectomy were performed, with the intrahepatic Glisson's approach or classical procedure respectively.

Results:

1. Clinical data include: operation time, intraoperative blood loss, volume of blood transfusion, complications and mortality, postoperative liver function,long-term curative effect were collected and analysed.
2. Statistical method: groups t-test univariate/multivariate analysis, logistic regression analysis, mixed linear regression, Cox survival analysis were used.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with liver malignant or benign disease distributed in a segment, lobe or half liver, malignant tumor ≤5 cm, without rupture, bleeding, and liver metastases, benign tumor ≤15cm.
2. Liver function > Child-pugh level B, no severe biliary cirrhosis, ICG ≤ 15%, the residual liver volume and standard liver volume ratio ≥ 40%. The conditions of open hepatectomy were achieved
3. Age: Between 18 to 70 years
4. Patients with regional stones distributed in a segment, lobe or half liver, combined or not combined with extrahepatic biliary calculi, hepatic parenchymal atrophy or fibrosis in the lesion region
5. Patients with good general condition, the conditions of open Anatomical Hepatectomy were achieved
6. Other organ lesions and previous biliary tract operation is not the absolute exclusion criteria
7. Written informed consent

Exclusion Criteria:

1. Patients with bad general condition or important organ lesions, liver resection could not be tolerated
2. Age:Younger than 18 or more than 70 years old
3. Malignant tumor recurrence within one month postoperation
4. Combined with severe liver atrophy hypertrophy syndrome, hepatic portal transposition or hilar biliary fibrosis / stenosis
5. Complicated case need to get emergency operation
6. Contraindication of laparoscopy: Combined with complicated acute cholangitis, repeated biliary tract operation, heavy intra-abdominal adhesion, Trocar can not be placed in. Artificial pneumoperitoneum could not be tolerated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with operation complication | Duration hospitalization(an expected average of 8 days)
  Operation time, intraoperative blood loss, volume of blood transfusion, complications and mortality, postoperative liver function were collected and analysed to evaluate the safety of the operation.

SECONDARY OUTCOMES:
Number of participants with abnormal liver function or discomfort symptoms induced by the operation | up to 3 years postoperation
  Liver function, quality of life and survival time were collected and analysed to evaluate the postoperative curative effect. The examination of ultrasound , CT and/or MR were perfomed in outpatient if necessary. The follow up interval time: every six months.

CONTACTS AND LOCATIONS:
Overall Officials: Shuguo Zheng, Study Director — Shuguo Zheng, MD Study Director Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Topal B, Aerts R, Penninckx F. Laparoscopic intrahepatic Glissonian approach for right hepatectomy is safe, simple, and reproducible. Surg Endosc. 2007 Nov;21(11):2111. doi: 10.1007/s00464-007-9303-z. Epub 2007 May 4. PMID 17479334
- [Background] Cho A, Asano T, Yamamoto H, Nagata M, Takiguchi N, Kainuma O, Souda H, Gunji H, Miyazaki A, Nojima H, Ikeda A, Matsumoto I, Ryu M, Makino H, Okazumi S. Laparoscopy-assisted hepatic lobectomy using hilar Glissonean pedicle transection. Surg Endosc. 2007 Aug;21(8):1466-8. doi: 10.1007/s00464-007-9253-5. Epub 2007 Mar 14. PMID 17356935
- [Background] Cho A, Yamamoto H, Kainuma O, Souda H, Ikeda A, Takiguchi N, Nagata M. Safe and feasible extrahepatic Glissonean access in laparoscopic anatomical liver resection. Surg Endosc. 2011 Apr;25(4):1333-6. doi: 10.1007/s00464-010-1358-6. Epub 2010 Sep 25. PMID 20872017
- [Background] Astudillo JA, Sporn E, Serrano B, Astudillo R. Ascariasis in the hepatobiliary system: laparoscopic management. J Am Coll Surg. 2008 Oct;207(4):527-32. doi: 10.1016/j.jamcollsurg.2008.05.020. Epub 2008 Jul 14. PMID 18926454
- [Background] Lai EC, Tang CN, Ha JP, Li MK. Laparoscopic liver resection for hepatocellular carcinoma: ten-year experience in a single center. Arch Surg. 2009 Feb;144(2):143-7; discussion 148. doi: 10.1001/archsurg.2008.536. PMID 19221325
- [Background] Dagher I, Diop PS, Lainas P, Carloni A, Franco D. Laparoscopic liver resection for localized primary intrahepatic bile duct dilatation. Am J Surg. 2010 Jan;199(1):131-5. doi: 10.1016/j.amjsurg.2008.12.027. Epub 2009 Apr 17. PMID 19375067
- [Background] Gigot JF, Hubert C, Banice R, Kendrick ML. Laparoscopic management of benign liver diseases: where are we? HPB (Oxford). 2004;6(4):197-212. doi: 10.1080/13651820410023950. PMID 18333077
- [Background] Koffron AJ, Stein JA. Laparoscopic liver surgery: parenchymal transection using saline-enhanced electrosurgery. HPB (Oxford). 2008;10(4):225-8. doi: 10.1080/13651820802166864. PMID 18773098
- [Background] Gumbs AA, Gayet B, Gagner M. Laparoscopic liver resection: when to use the laparoscopic stapler device. HPB (Oxford). 2008;10(4):296-303. doi: 10.1080/13651820802166773. PMID 18773113
- [Background] Belli G, Fantini C, D'Agostino A, Belli A, Russolillo N. Laparoscopic liver resections for hepatocellular carcinoma (HCC) in cirrhotic patients. HPB (Oxford). 2004;6(4):236-46. doi: 10.1080/13651820410023941. PMID 18333081
- [Background] Nguyen KT, Gamblin TC, Geller DA. World review of laparoscopic liver resection-2,804 patients. Ann Surg. 2009 Nov;250(5):831-41. doi: 10.1097/SLA.0b013e3181b0c4df. PMID 19801936
- [Derived] Liao KX, Yu F, Cao L, Wang BL, Li XS, Wang XJ, Li JW, Fan YD, Chen J, Zheng SG. Laparoscopic Glissonian pedicle versus hilar dissection approach hemihepatectomy: A prospective, randomized controlled trial. J Hepatobiliary Pancreat Sci. 2022 Jun;29(6):629-640. doi: 10.1002/jhbp.1129. Epub 2022 Mar 10. PMID 35224875